CLINICAL TRIAL: NCT06420518
Title: A Phase I Clinical Trial Testing the Accuracy of a Continuous Ketone Monitoring (CKM) System in Individuals With Type 1 Diabetes on Insulin Pump Therapy.
Brief Title: Accuracy of a Continuous Ketone Monitoring (CKM) System in Individuals With Type 1 Diabetes on Insulin Pump Therapy.
Acronym: CKM 1
Status: Completed | Type: Observational
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Melissa Rosina-Pasqua, Endocrinologist, McGill University Health Centre, Hygea Clinic, McGill University
Other Study IDs: 2024-10140
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: type1diabetes
Keywords: Continuous ketone monitoring system; Ketone monitoring; Diabetes ketoacidosis; diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Diet, Ketogenic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Continuous ketone monitoring (CKM) system: All study participants will wear the CKM system for the 2-week study duration. This timeframe is overlapped with both the outpatient phase (sequential ketogenic diets) and, inpatient phase (insulin-suspension period) of the study. The accuracy of the ketone values from the CKM will be assessed using standard point-of-care capillary ketone measurements as reference (control).
  Interventions: Other: Ketogenic diets; Other: 8-hour insulin-suspension period
- Standard point-of-care capillary ketone meter: All study participants will be asked to measure their ketone levels with a standard point-of-care capillary ketone meter once upon waking, before a meal and, 2-hours post-meal for the entire 2-week study duration. These ketone measurements will be used as reference values (control) for comparison with the readings from the CKM.
  Interventions: Other: Ketogenic diets; Other: 8-hour insulin-suspension period

INTERVENTIONS:
Other: Ketogenic diets — During the outpatient phase of the study, all participants will undergo a very low-carbohydrate diet (less than 50grams/day) and, a fasting diet (12 hours) in a randomized order. Both diets are 6 days in duration and, will be interspaced by an inpatient insulin-suspension period. These ketogenic diets are implemented to drive higher ketone levels, within a safe threshold, to assess the accuracy of the CKM sensor. All the while, study participants will be wearing the CKM and, taking multiple daily ketone measurements with a standard point-of-cate ketone meter.
Other: 8-hour insulin-suspension period — Interspaced between both ketogenic diets, on day 8 of the study, participants will have their insulin pumps suspended for 8 hours; therefore, participants will not receive any basal or bolus insulin. Ketone levels will be monitored on-site every 30 minutes with standard point-of-care capillary ketone meters and, if ketones measurements exceed the safety threshold, participants will be treated accordingly. Clearly defined stopping criteria and corrective treatments have been outlined in the study protocol to ensure participants safety.

SUMMARY:
The goal of this 14-day randomized pilot trial is to assess the accuracy of a continuous ketone monitoring (CKM) system when compared to standard point-of-care capillary ketone monitors in individuals with type 1 diabetes on insulin pump therapy. The main question it aims to answer is:

- Can a CKM system demonstrate equivalent ketone monitoring compared to a capillary ketone monitor with accuracy within a mean absolute difference of no more than ± 0.1 mmol/L.

Participants will be asked to wear the SiBio KS1 CKM system for 14-days while undergoing two sequential ketogenic diets which are interspaced by an inpatient insulin-suspension period.

DETAILED DESCRIPTION:
In this study, all study participants will wear the CKM system and collect multiple standard point-of-care capillary ketone measurements. Therefore, there will be two groups in terms of measurements methods, one acting as an active comparator (the CKM system) and, the other serving as a control (point-of-care capillary ketone measurements). Both groups of measurement methods will be assessed in all study participants for both the outpatient phase (sequential ketogenic diets) and, the inpatient phase (insulin-suspension period) of the study to evaluate the accuracy of the CKM system.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age.
2. A clinical diagnosis of type 1 diabetes (T1D) for at least one year, as per their treating diabetes physician in agreement with the primary investigator's clinical judgment (confirmatory C-peptide and antibodies will not be required).
3. On stable, commercial closed-loop pump therapy for the past 30 days.
4. Stable use of continuous glucose monitor system for the past 30 days.
5. Cellular phone with Android OS operating system 8.1 and above or iOS11 and above operating system, for data compatibility with continuous ketone monitor mobile app (SiCKM app).
6. Able to perform study related tasks.

Exclusion Criteria:

1. Current or ≤ 2 weeks use of sodium-glucose cotransporter-2 (SGLT2) inhibitor medication (e.g. empagliflozin).
2. Current use of ascorbic acid (Vitamin C) as it may impair accuracy of the sensor.
3. Severe hypoglycemic episode within one month of admission, defined as an event where glucose was <4 mmol/L resulting in seizure, loss of consciousness, needing third party assistance, or need to present to the emergency department.
4. Diabetic ketoacidosis episode requiring medical attention or intravenous insulin within one month.
5. Planned or ongoing pregnancy or breastfeeding individuals.
6. Any serious medical or psychiatric illness likely to interfere with ability to complete the trial, as per judgement of investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of this study are individuals with a type 1 diabetes diagnosis exceeding 1 year, using insulin pump therapy for more than one month. Participant recruitment for the study will predominantly occur through the Hygea Medical Clinic, complemented by outreach to previous study participants who have consented to future contact for research opportunities.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Overall MAD of ketone concentration of the CKM (active device) compared to ketone capillary-measurements (control) during the 8-hour insulin-suspension study. | 2 weeks

SECONDARY OUTCOMES:
Overall mean absolute difference (MAD) of ketone CKM (active device) concentration compared to ketone capillary-measurements at home (control). | 2 weeks
Mean difference (MD) of ketone CKM concentration compared to ketone capillary-measurements during the 8h insulin-suspension study. | 2 weeks
MD of ketone CKM concentration compared to ketone capillary-measurements at home. | 2 weeks
MAD & MD according to duration during outpatient period: | 2 weeks
  i)During the overall study period, ii) In the first 2 days of sensor life, iii)In the 13-14 days (last 2 days) of sensor life
MAD & MD across ketone levels during insulin-suspension visit: | 2 weeks
  i) ≥1.0, ii) ≥0.6, iii) ≤0.6
Number of participants experiencing ketones by both the CKM and capillary-ketone meter. | 2 weeks
  i) ≥0.6 during overall study period, inpatient period, outpatient period, ii) ≥1.0 during overall study period, inpatient period, outpatient period, iii) ≥1.5 mmol/L during overall study period, inpatient period, outpatient period
Glycemic and insulin outcomes will be compared between the very low-carbohydrate diet and the intermittent fasting diet. | 2 weeks
  i) Between 3.9 and 7.8 mmol/L, ii) Below 3.9 mmol/L and 3.0 mmol/L, iii) Above 10.0 mmol/L and 13.9 mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Melissa-Rosina Pasqua, MD, Principal Investigator — Hygea Medical Clinic
Locations (1):
- Hygea Clinic, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
The raw data (that is, insulin delivery, glucose levels and individual participant data) and informed consent form will be shared by the corresponding author, for academic purposes, subject to a material transfer agreement and approval of the McGill University Health Center's Research Ethics Board. All data shared will be de-identified. Raw data will be shared for non-commercial use upon reasonable request and a material transfer agreement.
Supporting Information: ICF